CLINICAL TRIAL: NCT03827434
Title: Improving Glycemic Control and Clinical Outcomes in Insulin Treated DM2 Patients Managed with CGM Devices and Clarity, a Randomized Clinical Trial
Brief Title: CGM/Clarity Use, Glycemic Control and Clinical Outcomes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We did not receive funding to conduct the study
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Baltimore VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ilias Spanakis, Assistant Professor of Medicine, VA Staff Physician, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00084458
Record Dates: First submitted 2019-01-28; First posted 2019-02-01 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus; Hyperglycemia; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia; Hypoglycemia | interventions — Point-of-Care Systems; Blood Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Continuous glucose Monitoring and Clarity (Active Comparator): Patients with DM2 and abnormal glycemic control followed by Continuous glucose Monitoring, using Clarity software
  Interventions: Device: Continuous glucose Monitoring Devices and Clarity Software
- Point of Care Fingerstick Glucose values (Placebo Comparator): Patients with DM2 and abnormal glycemic control followed by Point of Care Fingerstick Glucose values
  Interventions: Other: Point of Care (POC) blood glucose

INTERVENTIONS:
Device: Continuous glucose Monitoring Devices and Clarity Software — Patients with DM2 at the intervention group will be managed by Continuous glucose Monitoring and Clarity software
  Arms: Continuous glucose Monitoring and Clarity
Other: Point of Care (POC) blood glucose — Testing Blood Glucose levels with Point of Care (POC) blood glucose
  Arms: Point of Care Fingerstick Glucose values

SUMMARY:
The prevalence of Diabetes Mellitus (DM) is rising and more than 30 million of Americans or 9.4% of the US population has DM. Several large scale randomized clinical trials have found that improved glycemic control reduces the development of complications in patients with DM. However intensive glucose management carries an increased risk of hypoglycemia, a condition that may lead to neurological damage and is associated with increased incidence of cardiovascular events and mortality.

Reducing uncontrolled hyperglycemia and hypoglycemia represents therefore an important objective, as may decrease the direct and indirect impact that diabetes has in our health care system. Achieving optimal glycemic control requires frequent blood glucose monitoring by the patients and recurrent clinic visits,which is often difficult to achieve, as access to typical DM clinic is at least sub optimal.

m-Health and telemedicine health solutions represent alternative ways to manage patients in the outpatient setting and have been applied in different medical areas, among them in diabetes. However, almost all the telemedicine studies that have been previously performed and recruited DM patients used telemedicine solutions which were based on point of care (POC) finger-stick glucose testing, which are checked infrequently , usually 4-6 times/day.

Continuous glucose monitoring (CGM) devices offer additional ways to monitor blood glucose values and can provide numerous glucose measurements (as frequent as every 5 min). By using software applications, such as the Clarity (Dexcom), which highlights glucose patterns, trends and statistics in standardized reports, providers can make safe recommendations of adjusting DM medications, especially insulin titration. In this randomized clinical trial investigators propose to use CGM devices and Clarity software as a telemedicine platform in order to improve glycemic control and improve health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* History of Diabetes Mellitus type 2 (DM2) on insulin
* Uncontrolled glycemic control [hyperglycemia defined as Hba1c≥9% in the last 3 months or clinically important hypoglycemia (any reported glucose values less than 54 mg/dl) or severe hypoglycemia (low glucose value that led to a severe event characterized by altered mental status and or physical status requiring assistance)]

Exclusion Criteria:

* Subjects that have a history of type 1 DM
* History of type 2 DM, not treated or required to be treated with basal/bolus insulin (i.e diet only, any combination of non insulin antidiabetic drugs only, basal only insulin or bolus/short acting only insulin, or pre-mixed insulins) as these patients are less likely to benefit from CGM use.
* Pregnant patients
* Use of Clarity/ Share or follow applications as telehealth/telemedicine to improve DM management during the last 3 months prior to study entry.
* Extensive skin changes/disease or allergies that preclude wearing the CGM sensor
* Significant psychiatric illness or any mental condition rendering the subject incapable of understanding the objectives and potential consequences of the study.
* Subjects without personal computer and internet network access.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c (HbA1c) among participants who are managed with Continuous Glucose Monitoring Devices and Clarity versus participants who are managed with Point of Care glucose testing (standard of care) | Through study completion, 6 months after randomization
Change in the number of hypoglycemic episodes among participants who are managed with Continuous Glucose Monitoring Devices and Clarity versus participants who are managed with Point of Care glucose testing (standard of care) | Through study completion, 6 months after randomization
Change in the number of hospitalizations among participants who are managed with Continuous Glucose Monitoring Devices and Clarity versus participants who are managed with Point of Care glucose testing (standard of care) | Through study completion, 6 months after randomization
Change in the number of ED visits among participants who are managed with Continuous Glucose Monitoring Devices and Clarity versus participants who are managed with Point of Care glucose testing (standard of care) | Through study completion, 6 months after randomization
Change in mortality among participants who are managed with Continuous Glucose Monitoring Devices and Clarity versus participants who are managed with Point of Care glucose testing (standard of care) | Through study completion, 6 months after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Baltimore VA Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No, only de-identified data are going to be shared.